CLINICAL TRIAL: NCT04017754
Title: Low Plasma MBL Level is a Risk Factor for Recurrent Pregnancy Loss
Brief Title: Low Plasma Mannose Binding Lectin (p-MBL) Level is a Risk Factor for Recurrent Pregnancy Loss (RPL)
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Caroline Nørgaard-Pedersen, MD, Aalborg University Hospital
Other Study IDs: 36e19au5
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Results first posted 2021-02-24 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Recurrent Miscarriage; Spontaneous Abortion; Mannose-Binding Lectin Deficiency; Habitual Abortion; Pregnancy Complications; Pregnancy Loss; Recurrent Pregnancy Loss
Keywords: Mannose binding lectin; Perinatal outcome; Recurrent pregnancy loss
MeSH Terms: conditions — Abortion, Habitual; Abortion, Spontaneous; Mannose-Binding Protein Deficiency; Pregnancy Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples from the female patients and blood donors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study sample: In total, 267 women with unexplained recurrent pregnancy loss was included.
  Only patients with a history of 3 or more consecutive spontaneous pregnancy losses are included. Both biochemical and clinical losses documented in hospital records are accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social reasons are not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
- Reference Group: The MBL reference group comprised 185 Danish female blood donors of reproductive age (range 21 to 45 years), about whom we have no other information. After informed approval, all controls had an extra blood sample taken, which was analysed for p-MBL.

SUMMARY:
The present study is based on the hypothesis, that recurrent pregnancy loss (RPL) is associated with abnormal plasma mannose binding lectin (p-MBL) level. Secondarily, p-MBL level may affect the reproductive and the perinatal outcome in the first pregnancy following RPL. Thus, the present study aim to examine whether MBL should be a biomarker for women at risk for RPL and, secondarily, affect the reproductive and perinatal outcome, and thereby help clinicians identify fragile women who need intensified perinatal care.

DETAILED DESCRIPTION:
Recurrent pregnancy loss (RPL), defined as 3 or more consecutive pregnancy losses before 22 weeks of gestation, is a multifactorial disorder affecting 1-3% of all females of reproductive age. The underlying cause of RPL remain unknown in up to 50% of patients. Some of these patients may be affected by an aberrant immune system.

Low p-MBL levels have been associated with RPL, while relations to high p-MBL levels have been poorly studied. Reports concerning association between maternal p-MBL levels and perinatal outcomes including birth weight and gestational age are conflicting. Low p-MBL level may possess a negative effect by promoting an unfavorable immune response against foreign cells such as fetal/trophoblast cells.

This study is a single center a combined cross-sectional and prospective cohort study, that aims to investigate wether high and/or low p-MBL levels are associated with RPL (primary outcome) and whether it affects reproductive outcome in the first pregnancy following admission and the perinatal outcome in the first birth before and after admission (secondary outcome). If such associations exist, p-MBL could become an biomarker for the early identification of women with need for intensified perinatal care.

The study sample consists of Danish women admitted to the Centre for Recurrent Pregnancy Loss of Western Denmark. The study group includes 267 women with RPL. P-MBL levels in patients are compared to those of 185 female blood donors of fertile age with unknown reproductive history. The association between low p-MBL level and successful reproductive outcomes is analyzed with logistic regression adjusted for confounding variables (age, BMI and smoking). The perinatal outcomes in first birth (>22 weeks of gestation) before and after admission are compared between RPL subgroups according to their p-MBL level; low (≤500 ug/l), intermediate (501-3000 ug/l), and high (>3000 ug/l) p-MBL levels.

Female patients in the study group will have a blood sample taken at their first meeting in the the Centre for Recurrent Pregnancy Loss of Western Denmark before they become pregnant, and they will be followed until delivery of the first child after RPL, if pregnancy after RPL is achieved, or until end of study March 2021. Data on perinatal outcomes of pregnancies before and after RPL were collected at the first consultation, from hospital records, and, when needed, completed by telephone or e-mail correspondence.

ELIGIBILITY:
Inclusion Criteria:

- Women admitted to the Centre for Recurrent Pregnancy Loss of Western Denmark January 2016 to March 2020

Exclusion Criteria:

* Less than 3 consecutive pregnancy losses
* Significant uterine malformation on hydrosonography or hysteroscopy
* Significant chromosomal abnormalities
* Abnormal menstrual cycle length (<22 or >35 days) or irregular cycle
* Pregnancy at first meeting in the Recurrent Miscarriage Clinic
* Age <18 and >45 years

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female women of reproductive age.
Study Population: Women fulfilling the eligibility criteria will have p-MBL level measured from a blood sample when first admitted to the Centre for Recurrent Pregnancy Loss of Western Denmark and will be followed until delivery of the first child following the consecutive pregnancy losses, if pregnancy is achieved during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 452 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Nørgaard-Pedersen, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Norgaard-Pedersen C, Rom LH, Steffensen R, Kesmodel US, Christiansen OB. Plasma level of mannose-binding lectin is associated with the risk of recurrent pregnancy loss but not pregnancy outcome after the diagnosis. Hum Reprod Open. 2022 Jun 7;2022(3):hoac024. doi: 10.1093/hropen/hoac024. eCollection 2022. PMID 35747402

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study sample consisted of 267 female patients with RPL fulfilling the inclusion criterias.
Groups:
- Study Sample: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and additionally a parental chromosomal analysis in most cases.
- Control Group 1: The MBL control group comprised 185 Danish female blood donors of reproductive age (range 21 to 45 years), about whom we have no other information than their plasma MBL level. After informed approval, all controls had an extra blood sample taken, which was analysed for MBL.
Period: Overall Study
Arm/Group | Study Sample | Control Group 1
Started | 267 | 185
Completed | 267 | 185
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Sample: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
Arm/Group | Study Sample
Number analyzed (Participants) | 267
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 267
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 267
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 267
  Unknown | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 267
Body mass index [Mean (Full Range); unit: kg/m²] | 25.4 [16.8 to 50.0]
Number of consecutive pregnancy losses [Median (Full Range); unit: consecutive pregnancy losses] | 3 [3 to 13]
Percentage with primary Recurrent pregnancy loss (RPL) [Number; unit: Percentage of all RPL patients] | 53.9

OUTCOME MEASURES:

1. Primary Outcome: Plasma MBL Level (ug/ml)
Description: Manose Binding Lectin level in a blood sample
Time Frame: At first consultation. Results accessible within 3 weeks.
Population: 18 women were pregnant <12 weeks when blood sample was collected.
Measure: Median (Inter-Quartile Range); unit: ug/l
Groups:
- MBL Reference Group: The MBL reference group comprised 185 Danish female blood donors of reproductive age (range 21 to 45 years), about whom we have no other information than their plasma MBL level. After informed approval, all controls had an extra blood sample taken, which was analysed for MBL.
Arm/Group | Study Sample | MBL Reference Group
Number analyzed (Participants) | 267 | 185
ug/l | 717 [164 to 2131] | 1717 [505 to 3528]
Statistical Analysis 1: Comparison: Study Sample vs MBL Reference Group; Comparing the risk of low p-MBL level between RPL patients and MBL reference group. We hypothesized that more RPL patients had a low p-MBL level; thus, the null hypothesis was that no difference existed; Test type: Equivalence — A p-value <0.05 was considered significant for at difference in frequency of low p-MBL level(<500 ug/l) between groups; p < 0.001, Chi-squared; Prevalence proportion ratio = 1.79, 95% CI 2-sided [1.34 to 2.38] — The numerator is the risk of low p-MBL in the study sample with RPL patients and the denominator is the risk of low p-MBL in control group 1 of female blood donors

2. Secondary Outcome: Participants Giving Birth After Recurrent Pregnancy Loss (RPL) to a Child With Low Birth Weight
Description: <2500g
Time Frame: at delivery
Population: Patients who have given birth after admission within each p-MBL level subgroup
Measure: Number; unit: participants
Groups:
- RPL Patients With pMBL <500 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  79 RPL patients with p-MBL <500 ug/l gave birth after RPL, but birth weight was missing in 3 patients.
- RPL Patients With p-MBL >3000 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  23 RPL patients with p-MBL >3000 ug/l gave birth after RPL, but birth weight was missing in 2 patients.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 76 | 21
participants | 3 | 1

3. Secondary Outcome: Participants Giving Birth Before RPL to a Child With Low Birth Weight
Description: <2500g
Time Frame: At first consultation
Population: participants who had sRPL; thus, who had given birth before admission to at least one child. Data concerns first delivery.
Measure: Number; unit: participants
Groups:
- RPL Patients With pMBL <500 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  54 RPL patients with p-MBL <500 ug/l gave birth before RPL, but information on three of these births were excluded from this analysis since they were stillbirths.
- RPL Patients With p-MBL >3000 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  26 RPL patients with p-MBL >3000 ug/l gave birth before RPL but 1 was excluded from this analysis since it was a stillbirth.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 51 | 25
participants | 4 | 2

4. Secondary Outcome: Participants Giving Birth After RPL to a Child With Very Low Birth Weight
Description: <1500g
Time Frame: at delivery
Measure: Number; unit: participants
Groups:
- RPL Patients With pMBL <500 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  79 RPL patients with p-MBL <500 ug/l gave birth after RPL but birth weight was missing in 3 of these patients
- RPL Patients With p-MBL >3000 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  23 RPL patients with p-MBL >3000 ug/l gave birth after RPL, but birth weight was missing for 2 of these patients.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 76 | 21
participants | 0 | 0

5. Secondary Outcome: Participants Giving Birth Before RPL to a Child With Very Low Birth Weight
Description: <1500g
Time Frame: At first consultation
Measure: Count of Participants; unit: Participants
Groups:
- RPL Patients With pMBL <500 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  54 RPL patients with p-MBL <500 ug/l gave birth before RPL but information on three of these births were excluded from this analysis since they were stillbirths.
- RPL Patients With p-MBL >3000 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  26 RPL patients with p-MBL >3000 ug/l gave birth before RPL but information on one of these births were excluded from this analysis since it was a stillbirth.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 51 | 25
Participants | 0 | 0

6. Secondary Outcome: Participants With Preclampsia in Pregnancy After RPL
Description: High blood pressure and proteinuria
Time Frame: Developed from 20 weeks gestation and until 6 weeks postpartum. Data collected at delivery.
Measure: Count of Participants; unit: Participants
Groups:
- RPL Patients With pMBL <500 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  79 RPL patients with p-MBL <500 ug/l gave birth after RPL.
- RPL Patients With p-MBL >3000 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  23 RPL patients with p-MBL >3000 ug/l gave birth after RPL.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 79 | 23
Participants | 7 | 0

7. Secondary Outcome: Participants With Preclampsia in Pregnancy Before RPL
Description: High blood pressure and proteinuria
Time Frame: Developed from 20 weeks gestation and until 6 weeks postpartum. Data collected at first consultation.
Measure: Count of Participants; unit: Participants
Groups:
- RPL Patients With p-MBL >3000 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  26 RPL patients with p-MBL >3000 ug/l gave birth before RPL but information on one of these births were excluded from this analysis since was a stillbirth.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 51 | 25
Participants | 6 | 2

8. Secondary Outcome: Patients With Emergency Caesarean Section After RPL
Description: A surgical delivery in women who were planned for vaginal delivery initially, but an acute indication for caesarean delivery has since developed.
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Groups:
- RPL Patients With p-MBL >3000 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  23 RPL patients with p-MBL >3000 ug/l gave birth after RPL but 1 delivery method was missing.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 79 | 22
Participants | 10 | 4

9. Secondary Outcome: Patients With Emergency Caesarean Section Before RPL
Description: as for outcome 8
Time Frame: At first consultation
Measure: Count of Participants; unit: Participants
Groups:
- RPL Patients With pMBL <500 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  54 RPL patients with p-MBL <500 ug/l gave birth before RPL and data on one delivery method is missing.
- RPL Patients With p-MBL >3000 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  26 RPL patients with p-MBL >3000 ug/l gave birth before RPL but data on two delivery methods is missing.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 53 | 24
Participants | 12 | 6

10. Secondary Outcome: Patients With Elective Caesarean Section After RPL
Description: A surgical delivery in women who were planned for caesarean delivery
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Groups:
- RPL Patients With p-MBL >3000 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  23 RPL patients with p-MBL >3000 ug/l gave birth after RPL but data on one delivery method is missing.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 79 | 22
Participants | 13 | 3

11. Secondary Outcome: Patients With Elective Caesarean Section Before RPL
Description: A surgical delivery in women who were planned for caesarean delivery
Time Frame: At first consultation
Measure: Count of Participants; unit: Participants
Groups:
- RPL Patients With pMBL <500 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  54 RPL patients with p-MBL <500 ug/l gave birth before RPL but data on one delivery method is missing.
- RPL Patients With p-MBL >3000 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  26 RPL patients with p-MBL >3000 ug/l gave birth before RPL but data on two delivery methods were missing.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 53 | 24
Participants | 6 | 0

12. Secondary Outcome: Patients With Severe Peripartum Hemorrhage in Birth After RPL
Description: Hemorrhage of >999 ml
Time Frame: During delivery
Measure: Count of Participants; unit: Participants
Groups:
- RPL Patients With pMBL <500 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  79 RPL patients with p-MBL <500 ug/l gave birth after RPL but information on peripartum hemorrhage were missing in 1 case.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 78 | 23
Participants | 6 | 3

13. Secondary Outcome: Patients With Severe Peripartum Hemorrhage in Birth Before RPL
Description: Hemorrhage of >999 ml in minimum one previous birth befor RPL
Time Frame: At first consultation
Measure: Count of Participants; unit: Participants
Groups:
- RPL Patients With pMBL <500 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  54 RPL patients with p-MBL <500 ug/l gave birth before RPL but information on peripartum hemorrhage were missing for 9 patients.
- RPL Patients With p-MBL >3000 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  26 RPL patients with p-MBL >3000 ug/l gave birth before RPL but information on peripartum hemorrhage were missing for 5 patients.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 45 | 21
Participants | 8 | 0

14. Secondary Outcome: Patients With Moderate Peripartum Hemorrhage in Birth After RPL
Description: Hemorrhage of 500-1000 ml
Time Frame: During delivery
Measure: Count of Participants; unit: Participants
Groups:
- RPL Patients With pMBL <500 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  79 RPL patients with p-MBL <500 ug/l gave birth after RPL but data on one hemorrhage was missing.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 78 | 23
Participants | 21 | 2

15. Secondary Outcome: Patients With Moderate Peripartum Hemorrhage in Birth Before RPL
Description: Hemorrhage of 500-1000 ml in minumum one previous birth before RPL
Time Frame: At first consultation
Measure: Count of Participants; unit: Participants
Groups:
- RPL Patients With pMBL <500 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  54 RPL patients with p-MBL <500 ug/l gave birth before RPL but information on permpartum hemorrhage was missing for 9 patients.
- RPL Patients With p-MBL >3000 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  26 RPL patients with p-MBL >3000 ug/l gave birth before RPL but information on permpartum hemorrhage was missing for 5 patients.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 45 | 21
Participants | 6 | 6

16. Secondary Outcome: Patients With a Preterm Birth in Birth After RPL
Description: <37 weeks of gestation
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Groups:
- RPL Patients With pMBL <500 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  79 RPL patients with p-MBL <500 ug/l gave birth after RPL but information on gestational age was missing in 1 patient.
- RPL Patients With p-MBL >3000 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  23 RPL patients with p-MBL >3000 ug/l gave birth after RPL but information on gestational age was missing in 1 patient.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 78 | 22
Participants | 8 | 3

17. Secondary Outcome: Patients With a Preterm Birth in Birth Before RPL
Description: <37 weeks of gestation
Time Frame: At first consultation
Measure: Count of Participants; unit: Participants
Groups:
- RPL Patients With pMBL <500 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  54 RPL patients with p-MBL <500 ug/l gave birth before RPL, but information on 2 births were missing and 3 stillbirths were excluded.
- RPL Patients With p-MBL >3000 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  26 RPL patients with p-MBL >3000 ug/l gave birth before RPL but information on 2 births were missing and 1 stillbirth was excluded.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 49 | 23
Participants | 4 | 1

18. Secondary Outcome: Patients With a Very Preterm Birth in Birth After RPL
Description: <32 weeks of gestation
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Groups:
- RPL Patients With p-MBL >3000 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  23 RPL patients with p-MBL >3000 ug/l gave birth after RPL but information on gestational age was missing in 2 patients.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 78 | 21
Participants | 2 | 0

19. Secondary Outcome: Patients With a Very Preterm Birth in Birth Before RPL
Description: <32 weeks of gestation
Time Frame: At first consultation
Measure: Count of Participants; unit: Participants
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 49 | 23
Participants | 0 | 0

20. Secondary Outcome: Gender Ratio of Children Born After RPL
Description: Gender ratio in births before RPL
Time Frame: At delivery
Population: male:female ratio
Measure: Number; unit: male:female ratio
Groups:
- Study sampleRPL Patients With pMBL <500 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  79 RPL patients with p-MBL <500 ug/l gave birth after RPL. One of these births was a twin birth of same gender, which was counted as 1.
- RPL Patients With p-MBL >3000 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  23 RPL patients with p-MBL >3000 ug/l gave birth after RPL. One of these births was a twin birth of same gender, which was counted as 1.
Arm/Group | Study sampleRPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 79 | 23
male:female ratio | 1.08 | 2.29

21. Secondary Outcome: Gender Ratio of Children Born Before RPL
Description: Gender ratio in births after RPL
Time Frame: At first consultation
Measure: Number; unit: male:female ratio
Groups:
- RPL Patients With pMBL <500 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  54 RPL patients with p-MBL <500 ug/l gave birth before RPL and none of these were twins. 7 patients had >1 child birth before RPL of mixed gender and therefore excluded from this analysis.
- RPL Patients With p-MBL >3000 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  26 RPL patients with p-MBL >3000 ug/l gave birth before RPL and 3 patients had >1 child birth before RPL of mixed gender and therefore excluded from this analysis.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 47 | 23
male:female ratio | 3.27 | 1.88

22. Secondary Outcome: Patients With a Stillbirth After RPL
Description: Stillbirth are defined as fetal death >22 weeks of gestation and within 1 week after delivery
Time Frame: 1 week after delivery
Measure: Count of Participants; unit: Participants
Groups:
- RPL Patients With pMBL <500 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  67 RPL patients with p-MBL <500 ug/l gave birth after RPL.
- RPL Patients With p-MBL >3000 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  20 RPL patients with p-MBL >3000 ug/l gave birth after RPL.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 79 | 23
Participants | 0 | 0

23. Secondary Outcome: Patients With a Stillbirth Before RPL
Description: Stillbirth are defined as fetal death >22 weeks of gestation and within 1 week after delivery - all women with min one previous birth are included in this analysis.
Time Frame: At first consultation
Measure: Count of Participants; unit: Participants
Groups:
- RPL Patients With pMBL <500 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  54 RPL patients with p-MBL <500 ug/l gave birth >22 weeks before RPL.
- RPL Patients With p-MBL >3000 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  26 RPL patients with p-MBL >3000 ug/l gave birth >22 weeks before RPL.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 54 | 26
Participants | 4 | 3

24. Secondary Outcome: Patients With a Liveborn After RPL
Description: Number of women who give birth to a healthy liveborn child after RPL
Time Frame: Follow up at study end.
Measure: Count of Participants; unit: Participants
Groups:
- RPL Patients With pMBL <500 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  119 RPL patients had MBL>500 ug/l.
- RPL Patients With p-MBL >3000 ug/l: Women with unexplained recurrent pregnancy loss. Only patients with a history of 3 or more consecutive spontaneous pregnancy losses were included. Both biochemical and clinical losses documented in hospital records were accepted. Verified extrauterine pregnancy losses, complete molar pregnancies, and induced abortions of social and genetic reasons were not included in the total number of pregnancy losses. Women are excluded from this study, if they have significant uterine malformations, significant parental chromosomal abnormalities, irregular and/or abnormal length of their menstrual cycle length (<22 and >35 days interval), and/or no MBL measurement.
  At the first consultation in The Centre for Recurrent Pregnancy Loss of Western Denmark, all women have a diagnostic work-up, including collection of an obstetric and gynaecologic history, a routine blood analysis, a uterine hydrosonography, hysteroscopy, or hysterosalpingography, and a parental chromosomal analysis in most cases.
  46 patients had MBL>3000.
Arm/Group | RPL Patients With pMBL <500 ug/l | RPL Patients With p-MBL >3000 ug/l
Number analyzed (Participants) | 119 | 46
Participants | 79 | 23

ADVERSE EVENTS:
Time Frame: From January 2016 until March 2020 patients were admitted and serious adverse events were recorded from the day of admission to the RPL center and until birth (up to 2 years) or the end of the study in March 2020.
Description: Hospitalization due to abortion or birth was not considered as a serious adverse event.
  Only serious adverse events were recorded since no study specific intervention was performed.
Arm/Group | Study Sample
All-Cause Mortality (participants affected / at risk) | 0/267
Serious Adverse Events (participants affected / at risk) | 0/267
Other Adverse Events (participants affected / at risk) | 0/267

LIMITATIONS AND CAVEATS:
161 (60.3 %) patients gave birth after RPL during the study period, which limited the possibility to detect clear associations between p-MBL levels and perinatal outcomes after RPL.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT04017754/Prot_SAP_001.pdf